CLINICAL TRIAL: NCT06295484
Title: Effect of Nasal Continuous Positive Airway Pressure (nCPAP) Versus Non-Invasive Positive Pressure Ventilation (NIPPV) On Diaphragm Electrical Activity (Edi) In Very Low Birth Weight (VLBW) Preterm Infants
Brief Title: Effect of Nasal CPAP Versus NIPPV On Diaphragm Electrical Activity (Edi) In VLBW Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 5136
Record Dates: First submitted 2024-02-20; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Premature Lungs; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The baby will be assigned to first go on traditional CPAP, NIPPV, or high CPAP, stay for 2 hours, switch to one of the other methods for 2 hours and then spend 2 hours supported by the remaining method. We will continue to record the Edi signals during the 3 methods.
  Study duration will be 6 hours from the time of catheter insertion to fit into feeding and handling plans. Upon completion or termination of the study protocol, your baby will be put back to the originally prescribed breathing support.
  Routine monitoring for oxygen saturation, heart rate, and respiratory rate will be continued as per the standard of practice in the NICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Traditional CPAP, then NIPPV, then high CPAP. (Other): The participant will stay for 2 hours on Traditional CPAP, then 2 hours on NIPPV, then 2 hours on high CPAP. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP
- Traditional CPAP, then high CPAP, then NIPPV (Other): The participant will stay for 2 hours on Traditional CPAP, then 2 hours on high CPAP, then 2 hours on NIPPV. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP
- NIPPV, then traditional CPAP, then high CPAP (Other): The participant will stay for 2 hours on NIPPV, then 2 hours on traditional CPAP, then 2 hours on high CPAP. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP
- NIPPV, then high CPAP, then traditional CPAP. (Other): The participant will stay for 2 hours on NIPPV, then 2 hours on high CPAP, then 2 hours on traditional CPAP. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP
- High CPAP, then traditional CPAP, then NIPPV. (Other): The participant will stay for 2 hours on High CPAP, then 2 hours on traditional CPAP, then 2 hours on NIPPV. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP
- High CPAP, then NIPPV, then traditional CPAP. (Other): The participant will stay for 2 hours on High CPAP, then 2 hours on NIPPV, then 2 hours on traditional CPAP. The investigators will continue to record the Edi signals during the 3 methods.
  Interventions: Other: Alternating traditional CPAP, NIPPV, and high CPAP

INTERVENTIONS:
Other: Alternating traditional CPAP, NIPPV, and high CPAP — The investigators will continue to record the Edi signals during the 3 methods (traditional CPAP, NIPPV, and high CPAP)

SUMMARY:
Background:

In premature babies, many organ systems are not fully grown and developed, including the lungs and respiratory muscles, so they will need breathing support to help them to breathe by preventing their tiny air sacs to collapse. This support commonly done by CPAP and Non-Invasive Positive Pressure Ventilation (NIPPV) therapy by giving some pressure and oxygen to their lungs through an interface placed on their noses. Both (CPAP and NIPPV) can be used as a support modality for respiratory distress syndrome, apnea of prematurity, and providing breathing support after extubation from the full mechanical breathing support.

The CPAP supports the baby's immature lungs by delivering constant pressure to keep their lungs and breathing well supported. Whereas the NIPPV will use constant pressure in the background (similar to CPAP), and on top, it will give extra intermittent puffs at regular intervals to support the baby's breathing. The NIPPV is the most common choice by the clinicians when the traditional CPAP is no longer effective, to avoid the full mechanical breathing support and to protect the developing lungs.

Studies suggested that NIPPV is better than the traditional CPAP in reducing the need of the baby to need full mechanical breathing support. This might be because the investigators tend to use lower pressures with CPAP (5-8 cmH2O) compared to relatively higher pressures with NIPPV. More recently, clinicians showed the safety of using equivalent higher CPAP pressures (>9 cmH2O) to what the investigators use in the NIPPV in preterm babies.

One way to measure the support that the investigators are giving to the patient with the different devices is to measure the diaphragm activity, which the investigators call the Edi signal, using a special feeding catheter and a specific machine to measure it. The catheter is placed and used as a routine feeding tube but has sensors at the end to measure this Edi signal. One opening of the tube will be connected to a computer to record the Edi signals. The other opening of the tube will be used for feeding.

DETAILED DESCRIPTION:
Our main goal in this study:

To measure and compare the Edi in preterm babies requiring breathing support with CPAP or NIPPV.

Inclusion Criteria (Potential Candidates):

This study involves stable babies who were born with a birth weight of less than 1500 grams and require CPAP.

The steps of the study:

The baby will be assigned to first go on traditional CPAP, NIPPV, or high CPAP, stay for 2 hours, switch to one of the other methods for 2 hours and then spend 2 hours supported by the remaining method. The investigators will continue to record the Edi signals during the 3 methods.

Study duration will be 6 hours from the time of catheter insertion to fit into feeding and handling plans. Upon completion or termination of the study protocol, the participant's baby will be put back to the originally prescribed breathing support.

Routine monitoring for oxygen saturation, heart rate, and respiratory rate will be continued as per the standard of practice in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable preterm infants (defined as cardiovascular stability with normal blood pressure and heart rate for gestational age and no recent increase in apneic episodes or spells and confirmed by the attending neonatologist)
* Birth weight less than 1500 grams
* Admitted to the NICU at Sunnybrook Health Sciences Centre on nasal CPAP of 5 to 8 cmH2O support, for at least 48 hours and requiring less than 35% of oxygen

Exclusion Criteria:

* Congenital anomalies of the gastrointestinal tract
* Phrenic nerve damage
* Diaphragmatic paralysis
* Esophageal perforation
* Congenital or acquired neurological deficit (including significant intraventricular hemorrhage greater than Grade II) or neonatal seizure
* Significant congenital heart disease (including symptomatic PDA)
* Congenital anomalies of the diaphragm
* Congenital anomalies of the respiratory tracts (e.g., Congenital Cystic Adenomatoid Malformation 'CCAM')
* Ongoing treatment for sepsis
* Ongoing treatment for necrotizing enterocolitis (NEC)
* Ongoing treatment for lung infections
* Narcotic analgesics
* Gastric motility agents
* Infants on nasal CPAP and requiring more than 35% oxygen
* Infants with significant gastric residuals and vomiting
* Infants with facial anomalies
* Infants with pneumothorax or pneumomediastinum
* Infants in the immediate postoperative period

Ages: 1 Day to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The differences in Electrical Activity of the Diaphragm measured in MicroVoltage (Edi minimum) between: 1. Traditional CPAP versus NIPPV. 2. NIPPV versus CPAP (equivalent pressures in cmH2O). | 2 hours per each mode of ventilation, total of 6 hours Edi recording

SECONDARY OUTCOMES:
1. Neural respiratory rate per minute | 2 hours per each mode of ventilation, total of 6 hours
2. Edi peak measured in MicroVoltage | 2 hours per each mode of ventilation, total of 6 hours
3. The difference in transcutaneous pCO2 in mmHg | 2 hours per each mode of ventilation, total of 6 hours
4. The difference in oxygen requirements in percent (i.e, 21%) | 2 hours per each mode of ventilation, total of 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No